CLINICAL TRIAL: NCT05870462
Title: Semaglutide and Vascular Regeneration in People With Diabetes and/or Obesity
Brief Title: Semaglutide and Vascular Regeneration
Acronym: SEMA-VR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: Unity Health Toronto (Other); Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00068765
Record Dates: First submitted 2023-04-28; First posted 2023-05-23 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity
Keywords: GLP-1 receptor agonists; GLP-1; Semaglutide; Vascular regeneration; Inflammation; Monocytes; Granulocytes; Hematopoietic progenitor cells; Cardiovascular risk; Type 2 diabetes; Obesity
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity; Inflammation | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Participants will receive once-weekly semaglutide subcutaneous injection [Ozempic] at escalating doses from 0.25 mg/week, 0.5 mg/week, to 1.0 mg/week.
  Interventions: Drug: Semaglutide Pen Injector
- Usual care (No Intervention): Participants will continue to receive other usual medications, rehabilitation, procedures, and interventions as recommended by their healthcare providers.

INTERVENTIONS:
Drug: Semaglutide Pen Injector — * 0.25 mg/week (non-therapeutic dose) during Weeks 1-4
  * 0.50 mg/week during Weeks 5-8
  * 1.0 mg/week during Weeks 9-24
  Participants experiencing side effects (e.g. nausea, stomach pain, constipation, diarrhea, vomiting) at the maximum dose (1.0 mg/week) may be down-titrated to 0.50 mg/week.
  Participants who had been receiving a dipeptidyl peptidase 4 (DPP-4) inhibitor (sitagliptin, saxagliptin, linagliptin, alogliptin) will stop taking their DPP-4 inhibitor upon randomization to this arm.
  Other Names: Ozempic; Wegovy
  Arms: Semaglutide

SUMMARY:
SEMA-VR is a prospective, randomized, 6-month long, open-label study of semaglutide. Approximately 100 participants with type 2 diabetes and/or obesity will be randomized (1:1) to receive semaglutide at escalating doses (up to 1.0 mg/week) or usual care without semaglutide for 6 months.

The goal of this trial is to understand how semaglutide exerts cardio-protective effects in people with type 2 diabetes and/or obesity. The main question it aims to answer is:

• Does semaglutide treatment preserve or increase the number of vessel-repairing cells circulating in the blood?

Participants will:

* Be allocated to receive either semaglutide or usual care for 6 months
* Provide a blood sample at the baseline visit and another blood sample at the 6-month visit

Researchers will compare participants receiving semaglutide to those receiving usual care for any differences in the 6-month change in the number of vessel-repairing cells in the blood.

DETAILED DESCRIPTION:
The leading cause of death in people with type 2 diabetes (T2D) and/or obesity is atherosclerotic cardiovascular disease (ASCVD). Arterial damage and repair are regulated by mechanisms of vessel homeostasis, which include vasculogenesis (de novo blood vessel synthesis), angiogenesis (vessel formation from pre-existing vessels), and arteriogenesis (re-modelling of collateral vessels). Key cellular modulators of these processes include hematopoietic stem/progenitor cells (HPC) and their myeloid progenies, together referred to as vascular regenerative cells.

An established and innovative multi-parametric flow cytometry assay that utilizes lineage-specific cell surface marker expression and aldehyde dehydrogenase (ALDH) activity will be used to characterize and quantify vascular regenerative cells from peripheral blood samples. Using this assay, three distinct populations of vascular regenerative cells within the hematopoietic hierarchy have been previously identified:

* ALDHhiSSClow (high ALDH activity, low side scatter/granular complexity) represent primitive progenitor cells, such as HPCs, that secrete chemo-attractant cytokines to recruit other circulating vascular regenerative cells to sites of vessel damage and ischemia.
* ALDHhiSSCmid cells represent macrophage precursor cells (i.e. monocytes) classified along a spectrum of pro-inflammatory subtypes versus pro-vascular subtypes that remodel arterial occlusions.
* ALDHhiSSChi cells represent granulocyte precursors, consisting of a heterogeneous group of pro-inflammatory subtypes that aggravate atherosclerosis and endothelial damage, along with pro-angiogenic subtypes that reduce inflammation and support vessel repair.

Using this multi-parametric flow cytometry assay, it has been previously reported that people with T2D presented lower frequencies of vascular regenerative cells in their peripheral blood compared to people without T2D. In addition, these frequencies were increased in response to the antihyperglycemic agent empagliflozin and bariatric surgery, suggesting that this regenerative cell deficiency can be reversed. Specifically, three months after bariatric surgery, frequencies of ALDHhiSSClow primitive progenitor cells and pro-vascular ALDHhiSSCmid monocytes in the peripheral blood were increased, whereas frequencies of pro-inflammatory monocytes and ALDHhiSSChi granulocyte precursors were decreased. These studies established circulating vascular regenerative cells as key mechanistic constituents of vessel homeostasis that can be quantified from readily available blood samples, and highlighted the utility of the multi-parametric flow cytometry assay in providing high-throughput, real-time biological readouts of vascular repair potential or deficiency.

Semaglutide belongs to a drug class known as glucagon-like peptide-1 (GLP-1) receptor agonists (GLP-1RA). Semaglutide mimics the actions of GLP-1, a gut hormone that is released after a meal and triggers a range of metabotropic effects such as elevating insulin release, reducing food motility, and increasing satiety. In landmark clinical trials, weekly semaglutide injections led to a 1.9% reduction in HbA1c, 16% weight loss in adults and teens, and a 26% reduction in major ASCVD events.

The precise mechanism(s) underlying the effect of semaglutide on ASCVD reduction remain poorly defined. In light of previous observations (described above), the investigators hypothesize that in people with T2D, semaglutide add-on to usual care will be superior to usual care alone in the restoration of vascular regenerative cell frequency. Specifically, the investigators predict significantly greater baseline to 6 month increases in the frequency of ALDHhiSSClow primitive progenitor cells and pro-vascular ALDHhiSSCmid monocytes, along with decreases in pro-inflammatory monocytes and ALDHhiSSChi granulocyte precursors in the semaglutide-assigned group compared to the usual care group.

Findings from this study will reveal whether semaglutide affects the quantity of circulating vascular regenerative cells responsible for vessel repair, thereby providing a potential mechanism of action behind the reduction of ASCVD events observed in GLP-1RA cardiovascular outcome trials.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age who meet one of the following Health Canada indications to receive subcutaneous semaglutide injections:

   * Documented T2D with inadequate glycemic control
   * Body mass index (BMI) ≥ 30 kg/m^2 (obesity)
   * BMI ≥ 27 kg/m^2 (overweight) and at least one weight-related comorbidity, such as hypertension, dyslipidemia, or obstructive sleep apnea
2. AND meet one of the following ASCVD criteria:

   * History of ASCVD:

     * Documented coronary artery disease
     * Documented cerebrovascular or carotid disease
     * Documented peripheral artery disease
   * No ASCVD but has 2 or more of the following risk factors:

     * Cigarette smoker or stopped smoking within 3 months of screening
     * Persistent hypertension (defined as office blood pressure ≥ 140/90 mmHg) or currently on antihypertensive medications
     * BMI ≥ 27 kg/m^2
     * estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73m^2
     * Treated or untreated dyslipidemia
     * Triglyceride ≥ 2.0 mmol/L
     * HDL-C ≤ 1.0 mmol/L for men or ≤ 1.3 mmol/L for women
     * High sensitivity C-reactive protein (hsCRP) ≥ 2.0 mg/L
     * Documented micro- or macro-albuminuria
     * Self-identified South Asian ethnicity

Exclusion Criteria:

* Female subjects who are pregnant, planning pregnancy, or breastfeeding
* HbA1c > 11.0 %
* Currently on a GLP-1RA or previously taken a GLP-1RA
* Personal or family history of medullary thyroid carcinoma
* Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* New York Heart Association class IV symptoms of heart failure
* Known history of severe liver disease (e.g. Child-Pugh Class B or C)
* White blood cell count ≥ 15 x 10^9/L
* Active infectious disease requiring antibiotic or anti-viral agents
* Known acquired immunodeficiency syndrome such as HIV
* On oral steroid therapy (e.g. prednisone or other corticosteroids) or other immunosuppressive agents (e.g. methotrexate)
* Any malignancy not considered cured (except basal cell carcinoma of the skin). A subject is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening
* Any clinically significant or unstable medical condition that might limit one's ability to complete the study or comply with the requirements of the protocol, including: dermatologic disease, hematological disease, pulmonary disease, hepatic disease, gastrointestinal disease, genitourinary disease, endocrine disease, neurological disease, and psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the mean frequency (%) of circulating ALDHhiSSClow primitive progenitor cells in individuals treated with semaglutide versus usual care for 6 months | Baseline to 6 months post-randomization

SECONDARY OUTCOMES:
Changes in the mean frequency (%) of circulating ALDHhiSSCmid pro-vascular monocytes in individuals treated with semaglutide versus usual care for 6 months | Baseline to 6 months post-randomization
Changes in the frequency (%) of circulating ALDHhiSSCmid pro-inflammatory monocytes in individuals treated with semaglutide versus usual care for 6 months | Baseline to 6 months post-randomization
Changes in the frequency (%) of circulating ALDHhiSSChi pro-inflammatory granulocyte precursors in individuals treated with semaglutide versus usual care for 6 months | Baseline to 6 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — Unity Health Toronto; David A Hess, PhD, Principal Investigator — Robarts Research Institute, London, Ontario; David Mazer, MD, Study Chair — Unity Health Toronto; Hwee Teoh, PhD, Study Chair — Unity Health Toronto
Locations (2):
- Canada (2):
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hess DA, Verma S, Bhatt D, Bakbak E, Terenzi DC, Puar P, Cosentino F. Vascular repair and regeneration in cardiometabolic diseases. Eur Heart J. 2022 Feb 10;43(6):450-459. doi: 10.1093/eurheartj/ehab758. PMID 34849704
- [Background] Terenzi DC, Bakbak E, Trac JZ, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Isolation and characterization of circulating pro-vascular progenitor cell subsets from human whole blood samples. STAR Protoc. 2021 Feb 1;2(1):100311. doi: 10.1016/j.xpro.2021.100311. eCollection 2021 Mar 19. PMID 33554145
- [Background] Ghattas A, Griffiths HR, Devitt A, Lip GY, Shantsila E. Monocytes in coronary artery disease and atherosclerosis: where are we now? J Am Coll Cardiol. 2013 Oct 22;62(17):1541-51. doi: 10.1016/j.jacc.2013.07.043. Epub 2013 Aug 21. PMID 23973684
- [Background] Drucker DJ, Nauck MA. The incretin system: glucagon-like peptide-1 receptor agonists and dipeptidyl peptidase-4 inhibitors in type 2 diabetes. Lancet. 2006 Nov 11;368(9548):1696-705. doi: 10.1016/S0140-6736(06)69705-5. PMID 17098089
- [Result] Cappellari R, D'Anna M, Menegazzo L, Bonora BM, Albiero M, Avogaro A, Fadini GP. Diabetes mellitus impairs circulating proangiogenic granulocytes. Diabetologia. 2020 Sep;63(9):1872-1884. doi: 10.1007/s00125-020-05142-3. Epub 2020 Apr 18. PMID 32306097
- [Result] Terenzi DC, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Circulating Pro-Vascular Progenitor Cell Depletion During Type 2 Diabetes: Translational Insights Into the Prevention of Ischemic Complications in Diabetes. JACC Basic Transl Sci. 2018 Nov 5;4(1):98-112. doi: 10.1016/j.jacbts.2018.10.005. eCollection 2019 Feb. PMID 30847424
- [Result] Hess DA, Terenzi DC, Trac JZ, Quan A, Mason T, Al-Omran M, Bhatt DL, Dhingra N, Rotstein OD, Leiter LA, Zinman B, Sabongui S, Yan AT, Teoh H, Mazer CD, Connelly KA, Verma S. SGLT2 Inhibition with Empagliflozin Increases Circulating Provascular Progenitor Cells in People with Type 2 Diabetes Mellitus. Cell Metab. 2019 Oct 1;30(4):609-613. doi: 10.1016/j.cmet.2019.08.015. Epub 2019 Aug 30. PMID 31477497
- [Result] Hess DA, Trac JZ, Glazer SA, Terenzi DC, Quan A, Teoh H, Al-Omran M, Bhatt DL, Mazer CD, Rotstein OD, Verma S. Vascular Risk Reduction in Obesity through Reduced Granulocyte Burden and Improved Angiogenic Monocyte Content following Bariatric Surgery. Cell Rep Med. 2020 May 19;1(2):100018. doi: 10.1016/j.xcrm.2020.100018. eCollection 2020 May 19. PMID 33205058
- [Result] Sorli C, Harashima SI, Tsoukas GM, Unger J, Karsbol JD, Hansen T, Bain SC. Efficacy and safety of once-weekly semaglutide monotherapy versus placebo in patients with type 2 diabetes (SUSTAIN 1): a double-blind, randomised, placebo-controlled, parallel-group, multinational, multicentre phase 3a trial. Lancet Diabetes Endocrinol. 2017 Apr;5(4):251-260. doi: 10.1016/S2213-8587(17)30013-X. Epub 2017 Jan 17. PMID 28110911
- [Result] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Result] Sattar N, Lee MMY, Kristensen SL, Branch KRH, Del Prato S, Khurmi NS, Lam CSP, Lopes RD, McMurray JJV, Pratley RE, Rosenstock J, Gerstein HC. Cardiovascular, mortality, and kidney outcomes with GLP-1 receptor agonists in patients with type 2 diabetes: a systematic review and meta-analysis of randomised trials. Lancet Diabetes Endocrinol. 2021 Oct;9(10):653-662. doi: 10.1016/S2213-8587(21)00203-5. Epub 2021 Aug 20. PMID 34425083